CLINICAL TRIAL: NCT06588920
Title: Brain Activity, Cognitive Function, and Walking Ability in People With Parkinson's Disease
Brief Title: Brain Activity, Cognitive Function, and Walking Ability in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: NYCU113006AF1
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Older Adults; Parkinson Disease
Keywords: Executive function; Gait; Electroencephalography
MeSH Terms: conditions — Parkinson Disease | interventions — Gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease: People with Parkinson disease
  Interventions: Behavioral: Cognitive function, gait, and electroencephalogram
- Healthy older adults: Healthy older adults
  Interventions: Behavioral: Cognitive function, gait, and electroencephalogram

INTERVENTIONS:
Behavioral: Cognitive function, gait, and electroencephalogram — Measurement of cognitive function, gait performance, and electroencephalogram

SUMMARY:
The dual-task automated walking performance in people with Parkinson's disease (PD) is affected by their gait disturbances and impaired executive functions. Currently, the relationship between brain activity related to inhibitory control, executive functions, and dual-task walking performance in people with PD is not well understood. Therefore, this study aims to investigate the significance of different executive function domains on gait stability in healthy older adults and people with PD; whether brain activation related to inhibitory control is associated with gait stability in healthy older adults and people with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of idiopathic Parkinson disease
* Stable dopaminergic medicine ≥ 2 weeks
* Able to walk 10 meters without aid
* Mini-Mental Status Examination ≥ 24 points
* No uncorrected visual or auditory disorders
* Education at least junior high school
* No other disease may affect balance

Exclusion Criteria:

* Other medical diagnoses of neurological, musculoskeletal, or cardiopulmonary disorders
* History of brain surgery (e.g. deep brain stimulation)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital and community
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Gait variability | 1 day
  Using GAITRite system to measure the coefficient of variation (CV). The mean and standard deviation will be used to calculate the coefficient of variation (CV). CV = standard deviation / mean * 100%
Gait speed | 1 day
  Using GAITRite system to measure gait speed.
Step length | 1 day
  Using GAITRite system to measure step length
Step width | 1 day
  Using GAITRite system to measure step width.
Single support time | 1 day
  Using GAITRite system to measure single support time
Double support time | 1 day
  Using GAITRite system to measure double support time
Frontal Assessment Battery | 1 day
  The score ranged from 0 to 18. Higher scores show better executive function.
Trail making test | 1 day
  Trail making test contain part A and part B. Faster completing the test indicates better executive function.
Stroop color and word test | 1 day
  Record numbers of corrected color words which the subject responds within 45 sec.
Digit span test | 1 day
  Digit span test contain forward and backward part. Scores of forward digit span ranges from 0 to 16. Score of backward digit span ranges from 0 to 14. Higher scores indicate better executive function.
Event-related potential - N2 | 1 day
  Measure event-related potential through electroencephalography under single-task and dual-task paradigm.
Event-related potential - P300 | 1 day
  Measure event-related potential through electroencephalography under single-task and dual-task paradigm.
Go/Nogo test | 1 day
  Behavioral test during measuring electroencephalography.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan